CLINICAL TRIAL: NCT04157127
Title: Phase I Study of Th-1 Dendritic Cell Immunotherapy in Combination With Standard Chemotherapy for the Adjuvant Treatment of Pancreatic Adenocarcinoma (DECIST)
Brief Title: Th-1 Dendritic Cell Immunotherapy Plus Standard Chemotherapy for Pancreatic Adenocarcinoma
Acronym: DECIST
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Diakonos Oncology Corporation (Industry)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H-42434
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Adenocarcinoma; Pancreatic Cancer; Pancreatic Adenosquamous Carcinoma
Keywords: Immunotherapy; Adjuvant therapy; Cell Therapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label study where all subjects will receive the DC therapy. The number of cells administered will vary based on the group/cohort determination. Group A receives intervention after neoadjuvant chemotherapy, surgery and adjuvant chemotherapy. Group B contains 2 cohorts (low and high dose) with intervention (1st cycle) after surgery, but before adjuvant chemotherapy with the option for intervention after adjuvant chemotherapy (2nd cycle).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Autologous DC Therapy Group B Cohort 1 (Experimental): The DC therapy is manufactured from autologous dendritic cells loaded with tumor cell lysate and RNA. Patients will receive 2 doses of DC therapy (separated by 14 days) and be monitored (vital signs every 30 minutes) for 2 hours after each dose. During intervention, patients receive weekly peg-IFN at 180 mcg/week on the first day of administration up through 14 days after last dose.
  DC Therapy dose evaluated in Group B Cohort 1:
  First Cycle 1st dose - 8 million cells First Cycle 2nd dose - 8 million cells Second Cycle 1st dose - 8 million cells (optional) Second Cycle 2nd dose - 8 million cells (optional)
  Patients in Group B cohort 1 will receive the DC therapy after neoadjuvant chemotherapy and surgery (1st cycle), with an option for additional DC therapy (2nd cycle) after adjuvant chemotherapy.
  Interventions: Biological: Autologous DC Therapy
- Autologous DC Therapy Group B Cohort 2 (Experimental): The DC therapy is manufactured from autologous dendritic cells loaded with tumor cell lysate and RNA. Patients will receive 2 doses of DC therapy (separated by 14 days) and be monitored (vital signs every 30 minutes) for 2 hours after each dose. During intervention, patients receive weekly peg-IFN at 180 mcg/week on the first day of administration up through 14 days after last dose.
  DC Therapy dose evaluated in Group B Cohort 2:
  First Cycle 1st dose - 12 million cells First Cycle 2nd dose - 12 million cells Second Cycle 1st dose - 12 million cells (optional) Second Cycle 2nd dose - 12 million cells (optional)
  Patients in Group B cohort 2 will receive the DC therapy after neoadjuvant chemotherapy and surgery (1st cycle), with an option for additional DC therapy (2nd cycle) after adjuvant chemotherapy.
  Interventions: Biological: Autologous DC Therapy
- Autologous DC Therapy Group A (Experimental): ENROLLMENT IN THIS ARM HAS BEEN COMPLETED
  The DC therapy is manufactured from autologous dendritic cells loaded with autologous tumor cell lysate and mRNA. Patients will receive 3 doses of DC therapy (one every 14 days) and be monitored (vital signs every 30 minutes) for 2 hours after each dose. During intervention, patients receive weekly peg-IFN at 180 mcg/week on the first day of administration up through 14 days after last dose.
  DC Therapy dose evaluated in Group A:
  1. st dose - 0.5 million cells
  2. nd dose - 1 million cells
  3. rd dose - 2 million cells
  Patients in Group A will receive the DC therapy after neoadjuvant chemotherapy, surgery and adjuvant chemotherapy.
  Interventions: Biological: Autologous DC Therapy

INTERVENTIONS:
Biological: Autologous DC Therapy — Autologous DC Therapy

SUMMARY:
This is a phase 1, first in human, dose escalation study for safety and feasibility of multi-dose dendritic cell (DC) therapy for pancreatic ductal adenocarcinoma (PDAC) including adenosquamous carcinoma administered after surgical resection of PDAC.

DETAILED DESCRIPTION:
The primary objective of this phase 1, first in human trial is to determine the safety, toxicity, and feasibility of delivering autologous DCs loaded with pancreatic adenocarcinoma lysate and mRNA to pancreatic cancer patients following surgery.

After having undergone surgical resection of their PDAC (with or without prior neoadjuvant chemotherapy), patients will undergo apheresis for the manufacture of the DC therapy. Once the DC therapy has been manufactured, it will be administered by image-guided injections proximal to a lymph node near the surgical bed with concurrent use of subcutaneous peg-IFN. Patients will have the option to receive additional doses of the DC therapy and peg-IFN if they are eligible and interested.

ELIGIBILITY:
Inclusion Criteria

An individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Male or female, aged 18 years and older
3. Cytological or pathological confirmation of adenocarcinoma or adenosquamous carcinoma of the pancreas is deemed to be potentially resectable or borderline resectable based on tumor and host factors. This may include patients who undergo upfront resection or those who receive neoadjuvant chemotherapy +/- radiation prior to resection.
4. Adequate kidney, liver, bone marrow function, and immune function, as follows, within 28 days prior to registration:

   1. Hemoglobin ≥ 8.0 gm/dL
   2. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
   3. Platelet count ≥ 75,000 /mm3
   4. Total bilirubin ≤ 1.5 times upper limit of normal (ULN),
   5. Aspartate transaminase AST (SGOT) and alanine aminotransferase ALT (SGPT) ≤ 2.5 times the ULN
5. ECOG performance status ≤ 2.
6. For women of childbearing potential (WOCBP): use of highly effective contraception must be discussed with participants. NOTE: Patient must agree to start contraception at least 30 days before first vaccination and continue for at least 12 weeks after her last vaccination.
7. WOCBP must have a negative serum pregnancy prior to vaccination
8. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner during study participation and for an additional 12 weeks following discontinuations of last vaccination.
9. Patient must agree to not donate blood for up to 90 days after last vaccination.

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Unresectable or metastatic (stage IV) pancreatic cancer.
2. Patients with known HIV and a positive viral load.
3. Patients with active HBV and HCV infection. Those who are Hepatitis B sAb positive as well as those who are Hepatitis C Ab positive, but Hepatitis C RNA viral load negative will not be excluded.
4. Patients with any active autoimmune disease or immune deficiency or previous Guillain-Barre syndrome. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g. patient with psoriatic arthritis are excluded) are eligible provided all of the following conditions are met:

   1. Rash that covers less than 10 % of body surface area.
   2. Disease is well controlled at baseline and requires only low-potency topical corticosteroids.
   3. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
5. Use of nonstandard neoadjuvant chemotherapy regimen, as determined by the Investigator.
6. Female patients who are pregnant, breastfeeding, or of childbearing potential without a negative pregnancy test within 28 days (or decline contraception requirements as outlined above). Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
7. Patients unwilling or unable to comply with the protocol or provide informed consent.
8. Any severe or uncontrolled medical condition or other condition that could affect participation in this study (in the opinion of the investigator), including but not limited to hyper/hypothyroidism, active systemic autoimmune disorders, untreated viral hepatitis or autoimmune hepatitis.
9. Requires chronic treatment with a systemic steroid (⩾10 mg/day of prednisone equivalent) or with any systemic immunosuppressive agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety of DC Therapy | From treatment start until 6 weeks after.
  To determine the safety (measured by the frequency/duration of adverse events as defined by the Common Terminology Criteria for Adverse Events Version 5.0) and feasibility of delivering autologous dendritic cells loaded with pancreatic adenocarcinoma lysate and mRNA after surgical resection (evaluated by the ease of administering the study drug product proximal to a lymph node near the surgical bed).
Number of participants who experienced Dose Limiting Toxicities (DLTs) | From treatment start until 6 weeks after.
  A DLT is defined as any non-hematologic toxicity of grade 3 or 4 by the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE 5.0) that was probably or definitely DC-therapy related. Certain grade 4 hematologic toxicities that are probably or definitely DC-therapy related are also considered DLTs. Grade 2 or 3 myelosuppression that does not resolve or recover (with supportive measures) to grade 1 within 2 weeks that is probably or definitely DC-vaccine related is also considered a DLT. Grade 2 non-hematologic toxicities that do not resolve or recover (with supportive measures) to grade 1 within 2 weeks that are probably or definitely DC-therapy related are also considered DLTs. Any toxicity, regardless of grade, where systemic steroids are used as supportive care for management that is probably or definitely DC-therapy related is also considered a DLT.

SECONDARY OUTCOMES:
Recurrence-Free Survival | From surgery until recurrence or up to 3 years after surgery, whichever comes first.
  Measurement of time from resection surgery to recurrence of pancreatic adenocarcinoma.
Overall Survival | From surgery until death or up to 3 years after surgery, whichever comes first.
  Measurement of time from resection surgery to death.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Musher, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Baylor College of Medicine Medical Center - McNair Campus, Houston, Texas
  - Baylor St. Lukes Medical Center, Houston, Texas
  - Dan L. Duncan Cancer Center at Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.